CLINICAL TRIAL: NCT00551161
Title: An Open-label Exploratory Study With Memantine: Correlation Between Proton Magnetic Resonance Spectroscopy, Cerebrospinal Fluid Biomarkers, and Cognition in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Magnetic Resonance Spectroscopy Study of Memantine in Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Marc L Gordon, MD, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAM-MD-50
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; memantine; cholinesterase inhibitors; magnetic resonance spectroscopy; N-acetylaspartate; inositol; cerebrospinal fluid; tau proteins; amyloid beta-protein
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single-arm (Experimental): 24-week observational lead-in period, wherein patients already on a stable dose of donepezil, rivastigmine, or galantamine continue on that dose, followed by a 24-week open-label memantine period, wherein patients receive open-label memantine treatment titrated to a dose of 20 mg per day, in addition to their ongoing stable cholinesterase inhibitor treatment
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: memantine — 24-week observational lead-in period, wherein patients already on a stable dose of donepezil, rivastigmine, or galantamine continue on that dose, followed by a 24-week open-label memantine period, wherein patients receive open-label memantine treatment titrated to a dose of 10 mg orally b.i.d., in addition to their ongoing stable cholinesterase inhibitor treatment
  Other Names: Namenda

SUMMARY:
We are studying subjects with mild to moderate Alzheimer's disease who have been on a stable dose of any cholinesterase inhibitor [donepezil (Aricept), rivastigmine (Exelon), or galantamine (Razadyne)] for at least 3 months, and have not previously taken memantine (Namenda). This is an open-label study, with magnetic resonance spectroscopy (MRS) as the primary outcome measure, along with neuropsychological testing, and optional lumbar puncture, evaluating patients on their stable dose of a cholinesterase inhibitor over 24 weeks, followed by another 24 weeks on memantine in combination with stable dose of cholinesterase inhibitor. The purpose of this study is to characterize the progression of disease using MRS, cerebrospinal fluid (CSF) biomarkers, and cognitive outcome measures, and to determine whether changes in cognitive function on neuropsychological testing are correlated to changes in MR spectroscopic and/or CSF biomarkers.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia. The current US prevalence is estimated at over 4 million people, and it ranks as the 8th leading cause of mortality in the United States, accounting for over 60,000 deaths per year.

Memantine is the newest medication approved by the FDA for the treatment of AD. Since it works on a different transmitter system, it can be used in combination with the other FDA-approved treatments for AD, tacrine, donepezil, rivastigmine, or galantamine (collectively referred to as cholinesterase inhibitors).

It remains to be determined what effect currently available AD treatments have on the underlying structural and functional correlates of the dementia process. While preclinical evidence suggests that memantine decreases neuronal toxicity in vitro, it is not clear whether this translates into a beneficial effect in patients with AD.

One of the most pressing challenges underlying clinical trials in AD is the need to validate reliable surrogate biomarkers of disease progression. Proton magnetic resonance spectroscopy (MRS) allows for in vivo detection and measurement of brain metabolites. The spectroscopic features that have been most consistently observed in AD patients, as compared with patients with other causes of dementia, or with normal subjects, have been elevated myo-inositol (mI) and reduced N-acetylaspartate (NAA) .

Evaluation of cerebrospinal fluid (CSF) via lumbar puncture affords a minimally invasive window into the biochemical substrate enveloping the brain. Multiple previous studies of AD patients compared with control subjects have demonstrated decreased CSF beta-amyloid, and elevated CSF tau protein. Previous longitudinal studies have documented the stability of CSF beta-amyloid over one year and CSF tau over two years in AD, suggesting that these may be possible stable target measures for therapeutic intervention.

The purpose of this study is to characterize the progression of disease using MRS, CSF biomarkers, and cognitive outcome measures in patients with mild to moderate Alzheimer's disease after 24 weeks of observational treatment with stable dose of a cholinesterase inhibitor, and after another 24 weeks of open-label memantine treatment in addition to stable dose of a cholinesterase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from either the subject (if they have decisional capacity) or a Legally Authorized Representative (LAR) (as required by state or local law and the IRB), prior to the initiation of any study-specific procedures. (If a subject is unable to fully consent for himself/herself, but has capacity to appoint a research proxy, the legally authorized research proxy will be asked to sign consent, with the subject signing assent.)
* Male or female outpatients at least 50 years of age at Screening.
* If female, the patient must be at least two years postmenopausal or surgically sterile at Screening.
* The patient has a current diagnosis of probable Alzheimer's disease consistent with NINCDS-ADRDA criteria.
* The patient has a knowledgeable and reliable caregiver who will accompany the patient to all clinic visits during the course of the study.
* Mini-Mental State Examination (MMSE) score of at least 15 and not greater than 26 at Screening.
* Ongoing therapy with a stable dose of donepezil, rivastigmine, or galantamine for at least three months at the time of Screening.
* Physical examination, laboratory evaluations, and EKG results at Screening must be normal, or abnormal findings must be judged not clinically significant by the Investigator.
* The patient's MRI scan conducted as part of Screening (Visit 1) must be consistent with a diagnosis of Alzheimer's disease, and must not include any findings that could confound the spectroscopic analysis of subsequent MRIs (e.g., large cortical stroke, tumor, or other space-occupying brain lesions).
* Vision and hearing (hearing aid permissible) must be sufficient for compliance with testing procedures.
* The patient and/or their Legally Authorized Representative, and their caregiver must be able to speak, read, and understand English sufficiently to understand the nature of the study, to provide written informed consent, and to allow completion of all study assessments.

Exclusion Criteria:

* Clinically significant vitamin B12 deficiency at Screening.
* Patients with a modified Hachinski ischemia score greater than 4 at Screening.
* Patients with evidence of clinically significant and active pulmonary, gastrointestinal, renal, hepatic, endocrine, or cardiovascular system disease. Patients with controlled hypertension and right bundle branch block (complete or partial) may be included in the study. Patients with thyroid disease may also be included in the study provided they are euthyroid on treatment. Patients with controlled diabetes may also be included.
* Patients with severe renal impairment (estimated creatinine clearance < 35 mL/min).
* Patients with systolic blood pressure (while sitting) greater then than 180 mm Hg or less then 90 mm Hg, or diastolic blood pressure (while sitting) greater than 100 mm Hg or less than 50 mm Hg at Screening.
* Patients with evidence of other neurological disorders including, but not limited to, stroke, Parkinson's disease, seizure disorder, hydrocephalus, or head injury with loss of consciousness within the past five years at Screening.
* Patients with a current DSM-IV Axis I disorder other than Alzheimer's disease, including schizophrenia or schizoaffective disorder, bipolar disorder, current major depressive episode, psychosis, panic disorder, or post-traumatic stress disorder.
* Patients with dementia complicated by other organic disease.
* Patients who have had a previous brain scan (MRI or CT) with results inconsistent with a diagnosis of probable Alzheimer's disease.
* Patients with an oncological diagnosis (hematological or solid tumor) which is currently being treated, or for which there has been treatment within the year preceding Screening, or for which there is still evidence of active disease. (Note: Patients with local dermatological tumors at such as basal or squamous cell carcinoma may be included.)
* Patients with an object in the head or neck which would invalidate or obstruct the successful completion of an MRI scan, or patients who have other contraindications to MRI, including those with implanted ferromagnetic material or devices such as cardiac pacemakers, deep brain stimulators, cochlear implants, or intraocular metallic shards.
* Patients who are claustrophobic and/or unable to tolerate MRI at Screening, or whom the Investigator believes will not be able to tolerate further scans scheduled during the course of the study.
* Patients with a known or suspected history (within the past 5 years at Screening) of alcoholism or drug abuse.
* Patients who are on an unstable dose of a cholinesterase inhibitor (donepezil, rivastigmine, or galantamine), are currently taking more than one cholinesterase inhibitor at Screening, who are likely to require a change in cholinesterase drug dose during the course of the study, or for whom a cholinesterase inhibitor therapy is contraindicated.
* Patients with a history of severe drug allergy or hypersensitivity, or patients with known hypersensitivity to memantine, amantadine, rimantadine, or lactose.
* Patients who have been previously treated with or have participated in an investigational study of neramexane, memantine, or amantadine.
* Patients previously treated with commercial memantine.
* Patients who have been in an investigational drug study or who have received treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) of Screening.
* Patients or caregivers who are unwilling or unable to abide by the visit schedule and other requirements of the study.
* Any condition which would make the patient or caregiver unsuitable for the study in the opinion of the Investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Gordon, M.D., Principal Investigator — Northwell Health
Locations (1):
- The Litwin-Zucker Research Center, Manhasset, New York, United States

REFERENCES:
- [Background] Adalsteinsson E, Sullivan EV, Kleinhans N, Spielman DM, Pfefferbaum A. Longitudinal decline of the neuronal marker N-acetyl aspartate in Alzheimer's disease. Lancet. 2000 May 13;355(9216):1696-7. doi: 10.1016/s0140-6736(00)02246-7. PMID 10905250
- [Background] Anderson RN, Smith BL. Deaths: leading causes for 2002. Natl Vital Stat Rep. 2005 Mar 7;53(17):1-89. PMID 15786629
- [Background] Andreasen N, Hesse C, Davidsson P, Minthon L, Wallin A, Winblad B, Vanderstichele H, Vanmechelen E, Blennow K. Cerebrospinal fluid beta-amyloid(1-42) in Alzheimer disease: differences between early- and late-onset Alzheimer disease and stability during the course of disease. Arch Neurol. 1999 Jun;56(6):673-80. doi: 10.1001/archneur.56.6.673. PMID 10369305
- [Background] Benton A, Hannay HJ, Varney NR. Visual perception of line direction in patients with unilateral brain disease. Neurology. 1975 Oct;25(10):907-10. doi: 10.1212/wnl.25.10.907. PMID 1237101
- [Background] Buschke, H. Selective reminding for analysis of memory and learning. J Verb Learn and Verb Behav 12:543-550, 1975.
- [Background] Buschke H, Fuld PA. Evaluating storage, retention, and retrieval in disordered memory and learning. Neurology. 1974 Nov;24(11):1019-25. doi: 10.1212/wnl.24.11.1019. No abstract available. PMID 4473151
- [Background] Chen HS, Pellegrini JW, Aggarwal SK, Lei SZ, Warach S, Jensen FE, Lipton SA. Open-channel block of N-methyl-D-aspartate (NMDA) responses by memantine: therapeutic advantage against NMDA receptor-mediated neurotoxicity. J Neurosci. 1992 Nov;12(11):4427-36. doi: 10.1523/JNEUROSCI.12-11-04427.1992. PMID 1432103
- [Background] Cohen JR, Elvevag B, Goldberg TE. Cognitive control and semantics in schizophrenia: an integrated approach. Am J Psychiatry. 2005 Oct;162(10):1969-71. doi: 10.1176/appi.ajp.162.10.1969. PMID 16199848
- [Background] Dixon RM, Bradley KM, Budge MM, Styles P, Smith AD. Longitudinal quantitative proton magnetic resonance spectroscopy of the hippocampus in Alzheimer's disease. Brain. 2002 Oct;125(Pt 10):2332-41. doi: 10.1093/brain/awf226. PMID 12244089
- [Background] Frederick BD, Lyoo IK, Satlin A, Ahn KH, Kim MJ, Yurgelun-Todd DA, Cohen BM, Renshaw PF. In vivo proton magnetic resonance spectroscopy of the temporal lobe in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2004 Dec;28(8):1313-22. doi: 10.1016/j.pnpbp.2004.08.013. PMID 15588758
- [Background] Hamsher KD, Roberts RJ. Memory for recent U.S. presidents in patients with cerebral disease. J Clin Exp Neuropsychol. 1985 Feb;7(1):1-13. doi: 10.1080/01688638508401238. PMID 3980677
- [Background] Hoyert DL, Kung HC, Smith BL. Deaths: preliminary data for 2003. Natl Vital Stat Rep. 2005 Feb 28;53(15):1-48. PMID 15779680
- [Background] Huang W, Alexander GE, Chang L, Shetty HU, Krasuski JS, Rapoport SI, Schapiro MB. Brain metabolite concentration and dementia severity in Alzheimer's disease: a (1)H MRS study. Neurology. 2001 Aug 28;57(4):626-32. doi: 10.1212/wnl.57.4.626. PMID 11524470
- [Background] Jessen F, Traeber F, Freymann K, Maier W, Schild HH, Block W. Treatment monitoring and response prediction with proton MR spectroscopy in AD. Neurology. 2006 Aug 8;67(3):528-30. doi: 10.1212/01.wnl.0000228218.68451.31. PMID 16894124
- [Background] Keilhoff G, Wolf G. Memantine prevents quinolinic acid-induced hippocampal damage. Eur J Pharmacol. 1992 Sep 4;219(3):451-4. doi: 10.1016/0014-2999(92)90487-o. PMID 1425971
- [Background] Lin A, Ross BD, Harris K, Wong W. Efficacy of proton magnetic resonance spectroscopy in neurological diagnosis and neurotherapeutic decision making. NeuroRx. 2005 Apr;2(2):197-214. doi: 10.1602/neurorx.2.2.197. PMID 15897945
- [Background] Linker G, Mirza N, Manetti G, Meyer M, Putnam KT, Sunderland T. Fine-needle, negative-pressure lumbar puncture: a safe technique for collecting CSF. Neurology. 2002 Dec 24;59(12):2008-9. doi: 10.1212/01.wnl.0000038360.01635.39. No abstract available. PMID 12499507
- [Background] Miguel-Hidalgo JJ, Alvarez XA, Cacabelos R, Quack G. Neuroprotection by memantine against neurodegeneration induced by beta-amyloid(1-40). Brain Res. 2002 Dec 20;958(1):210-21. doi: 10.1016/s0006-8993(02)03731-9. PMID 12468047
- [Background] Modrego PJ, Fayed N, Pina MA. Conversion from mild cognitive impairment to probable Alzheimer's disease predicted by brain magnetic resonance spectroscopy. Am J Psychiatry. 2005 Apr;162(4):667-75. doi: 10.1176/appi.ajp.162.4.667. PMID 15800137
- [Background] Rose SE, de Zubicaray GI, Wang D, Galloway GJ, Chalk JB, Eagle SC, Semple J, Doddrell DM. A 1H MRS study of probable Alzheimer's disease and normal aging: implications for longitudinal monitoring of dementia progression. Magn Reson Imaging. 1999 Feb;17(2):291-9. doi: 10.1016/s0730-725x(98)00168-4. PMID 10215485
- [Background] Sunderland T, Wolozin B, Galasko D, Levy J, Dukoff R, Bahro M, Lasser R, Motter R, Lehtimaki T, Seubert P. Longitudinal stability of CSF tau levels in Alzheimer patients. Biol Psychiatry. 1999 Sep 15;46(6):750-5. doi: 10.1016/s0006-3223(99)00143-2. PMID 10494442
- [Background] Waldman AD, Rai GS. The relationship between cognitive impairment and in vivo metabolite ratios in patients with clinical Alzheimer's disease and vascular dementia: a proton magnetic resonance spectroscopy study. Neuroradiology. 2003 Aug;45(8):507-12. doi: 10.1007/s00234-003-1040-y. Epub 2003 Jul 22. PMID 12879326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August, 2007 through May, 2010, at the Litwin-Zucker Research Center
Groups:
- Memantine: 24-week observational lead-in period, wherein patients already on a stable dose of donepezil, rivastigmine, or galantamine continue on that dose, followed by a 24-week open-label memantine period, wherein patients receive open-label memantine treatment titrated to a dose of 20 mg per day, in addition to their ongoing stable cholinesterase inhibitor treatment
Period: Overall Study
Arm/Group | Memantine
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single-arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Metabolite Ratios of N-acetylaspartate (NAA) to Creatine (Cr), Myo-inositol (mI) to Cr, Choline (Cho) to Cr, NAA to Cho, and NAA to mI, on Cholinesterase Monotherapy vs Combination of Memantine and Cholinesterase Inhibitor
Description: Ratios of myo-inositol (mI), N-acetylaspartate (NAA), total creatine (Cr), and choline (Cho) by single voxel 1H MRS (proton magnetic resonance spectroscopy). Mean (± SD) metabolite levels (normalized to T2-corrected water signal intensity) and metabolite ratios for Alzheimer's disease subjects at baseline (t0), after 24 weeks of ongoing monotherapy with stable-dose cholinesterase inhibitor (t1), and after another 24 weeks of combination therapy with memantine in addition to stable-dose cholinesterase inhibitor (t2). The Wilcoxon signed-rank test was used to examine whether the change between t0 and t1 differed from the change between t1 and t2 [(t2 - t1) - (t1 - t0)].
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ratio (normalized to T2-corrected water
Arm/Group | Memantine
Number analyzed (Participants) | 11
ratio (normalized to T2-corrected water
  Change in NAA [(t2-t1) - (t1-t0)] | -54 (102)
  Change in Cr [(t2-t1) - (t1-t0)] | -2 (36)
  Change in Cho [(t2-t1) - (t1-t0)] | 9 (12)
  Change in mI [(t2-t1) - (t1-t0)] | 16 (23)
  Change in NAA/Cr [(t2-t1) - (t1-t0)] | -0.09 (0.15)
  Change in Cho/Cr [(t2-t1) - (t1-t0)] | 0.02 (0.06)
  Change in mI/Cr [(t2-t1) - (t1-t0)] | 0.04 (0.08)
  Change in NAA/Cho [(t2-t1) - (t1-t0)] | -0.26 (0.39)
  Change in NAA/mI [(t2-t1) - (t1-t0)] | -0.35 (0.50)
Statistical Analysis 1: Comparison: Memantine; The Wilcoxon signed-rank test was used to examine whether the change between t0 and t1 differed from the change between t1 and t2 [(t2 - t1) - (t1 - t0)] for each of the metabolites and ratios, in order to examine whether the rate of change differed while on monotherapy as compared with combination therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Due to the exploratory nature of these analyses, no adjustment for multiple testing was made. Although it would have been preferable to carry out an omnibus analysis, due to the small sample size, the descriptive approach described above was used

ADVERSE EVENTS:
Arm/Group | Single-arm
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No